CLINICAL TRIAL: NCT02723890
Title: The Efficacy and Safety of Using the Novel Tyto Device for Remote Physical Examination by a Physician as Compared to a Standard Medical Physical Examination
Brief Title: The Efficacy and Safety of Using the Novel Tyto Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, waisman yehezkel, Associate Professor, MD, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RMC-15-0266
Record Dates: First submitted 2016-03-01; First posted 2016-03-31 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Pharyngitis; Respiratory Diseases; Cardiac Diseases; Ear Infection
MeSH Terms: conditions — Pharyngitis; Respiratory Tract Diseases; Heart Diseases; Otitis

ARMS (1):
- Tyto Device (Experimental): examination with Tyto device carried out by a nurse and sent online to the principle and co-investigators for remote analysis.
  Interventions: Device: Tyto Device

INTERVENTIONS:
Device: Tyto Device

SUMMARY:
To investigate the efficacy and safety of using the novel Tyto device for remote physical examination by co-investigators as compared to a standard medical physical examination by physicians.

DETAILED DESCRIPTION:
A single center, prospective, qualitative study. Patients referred to the emergency department will be triaged according to The Canadian Triage & Acuity Scale (CTAS).

Patients presenting with complaints suitable for examination with the Tyto device (ear/throat/respiratory/cardiac complaints) and meeting the inclusion criteria will be informed and asked for consent. Patients participating in the study will be referred to a room dedicated for the purpose.

A minimum of a hundred volunteer patients will be selected and enrolled for a preliminary Pilot Study. Final study design and its extent will be determined accordingly.

Physical examinations using the Tyto device will be performed by the co-investigators, and sent online to the principle investigator for remote analysis.

The emergency department physician will examine the patient using conventional examination instruments (i.e. stethoscope, otoscope).

The data collected will be recorded on predetermined case report form (CRF), timed, stored and analyzed by the principle and co-investigators. The findings of the co-investigators' examination will be compared to the conventional examination instruments used by the emergency department physician.

Results will be checked and compared categorically (0-inconclusive; 1-normal; 2-pathological findings)

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to the Emergency department and are categorized between 2-5 on the Canadian Triage & Acuity Scale (CTAS) scoring scale.

Exclusion Criteria:

* CTAS 1.
* Pregnant adolescent.
* Multi-drug resistant carriers.
* Intellectual disability disorders.
* Unsigned informed consent.

  * Patients with CTAS score of 2-3, will be first addressed by a physician to ascertain their eligibility to be enrolled to the study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 136 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
The concordance of diagnosis and physical findings using the Tyto device on the heart, lung ear and throat as compared to standard physical examination (normal heart and lung sounds, arrhythmia, crackles, normal appearance of ear and throat or otherwise) | up to 6 hrs
  during the visit to the emergency department.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 6 hrs
  during the visit to the emergency department.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Emergency Medicine, Schneider Children's Medical Center of Israel, Petah Tikva, Israel